CLINICAL TRIAL: NCT03803163
Title: A Phase 1, Open-Label, Dose Escalation Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single Doses of TransCon PEG Treprostinil Administered as a Subcutaneous Injection in Healthy Adult Male Volunteers
Brief Title: A Safety, Tolerability and Pharmacokinetics Study of TransCon Treprostinil in Healthy Adult Male Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Discontinued early due to local tolerance expectations not being met.
Sponsor: Ascendis Pharma A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TCP-PH-101
Record Dates: First submitted 2019-01-10; First posted 2019-01-14 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TransCon Treprostinil (Experimental)
  Interventions: Drug: TransCon Treprostinil

INTERVENTIONS:
Drug: TransCon Treprostinil
  Other Names: ACP-009

SUMMARY:
To determine the maximum tolerated dose (MTD) and assess safety and tolerability of escalating single doses of TransCon PEG treprostinil administered as a subcutaneous injection to healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Subject gives voluntary written informed consent to participate in the study.
2. Subject is a healthy male between the ages of 18 and 50 years, inclusive, at Screening.
3. Subjects must weigh between 60 and 120 kg, inclusive, with a BMI between 19.0-32.0 kg/m2, inclusive at Screening.
4. Subject has a medical history, physical examination, vital signs, ECG and clinical laboratory results within normal limits or considered not clinically significant by the Investigator at Screening.
5. Subject agrees to abstain from taking any prescription medication for 14 days prior to check-in and to abstain from taking any non-prescription medications (except multivitamins) or herbal supplements for 7 3 days prior to check-in Baseline until discharge from the study (unless prescribed by the Investigator to treat an AE).
6. Subject agrees to abstain from consuming alcohol from three days prior to check-in and until discharge from the study.
7. Subject agrees to refrain from strenuous exercise from check-in and until discharge from the study.
8. Subject is able to communicate effectively with study personnel and be considered reliable, willing and cooperative in terms of compliance with the protocol requirements.

Exclusion Criteria:

1. Subject has any clinically relevant abnormality identified during the screening physical examination, 12-lead ECG, or laboratory examinations.
2. Subject has a history of anaphylaxis, a previous documented hypersensitivity reaction, or a clinically significant idiosyncratic reaction to any drug.
3. Subject has a clinically significant history of neurological, cardiovascular, respiratory, endocrine, hematological, hepatic, renal, gastrointestinal, genitourinary, pulmonary, and/or musculoskeletal disease; glaucoma; a psychiatric disorder, or any other chronic disease, whether controlled by medication or not.
4. Subject has a history of postural hypotension, or unexplained syncope.
5. Subject has a blood pressure that is less than 90 mmHg systolic or 50 mmHg diastolic at Screening or Baseline.
6. Subject has a pulse rate that is greater than 90 bpm after sitting at rest for at least 5 minutes at Screening or Baseline.
7. Subject has a history of hypertension.
8. Subject has a blood pressure that is greater than 150 mmHg systolic or 90 mmHg diastolic at Screening or Baseline
9. Subject has a predisposing condition that could interfere with the absorption, distribution, metabolism, or excretion of drugs.
10. Subject has tested positive at the screening visit for HIV infection, HBsAg, or the HCV antibody.
11. Subject currently uses tobacco or nicotine products or has a history of tobacco use within six months prior to Baseline.
12. Subject has a history of alcohol abuse or a history of or current impairment of organ function reasonably related to alcohol abuse.
13. Subject has a history of or current evidence of abuse of licit or illicit drugs, including a positive urine screen for drugs of abuse at Screening or Baseline.
14. Subject has a history of abnormal bleeding tendencies.
15. Subject has donated blood or plasma or has lost a significant volume of blood (greater than 450 mL) within four weeks prior to Baseline.
16. Subject has participated in any investigational drug study within 30 days prior to their initial Screening visit.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 42 days
  Safety and tolerability of single doses of TransCon Treprostinil treatment

SECONDARY OUTCOMES:
Maximum Plasma Concentration [Cmax] of TransCon Treprostinil | 42 days
  Pharmacokinetic profile of single doses of TransCon Treprostinil